CLINICAL TRIAL: NCT03184298
Title: Piloting ProHealth: A Program for Male Soldiers on Sex, Dating and Alcohol-Use at Fort Bragg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: Rhode Island Hospital (Other); University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RHC-A-18-011; W81XWH-15-2-0055 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Sexual Assault and Rape; Risk Behavior; Alcohol Abuse
Keywords: Military Personnel; Sexual Assault; Military Sexual Trauma; Alcohol and Substance Abuse
MeSH Terms: conditions — Risk-Taking; Alcoholism; Military Sexual Trauma; Substance-Related Disorders | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Other): Participants receive three interventions: Surveys, Interviews, and Group Workshops
  Interventions: Other: Surveys; Other: Interviews; Other: Group Discussions

INTERVENTIONS:
Other: Surveys — The purpose of the surveys is to collect quantitative data to determine the relative impact of the intervention program on participants' sexual behaviors and alcohol use.
Other: Interviews — These Motivational Interviews aim to promote change in behavior through open-ended questions, affirmations, and reflections.
Other: Group Discussions — The purpose of the group workshop is to create discussions surrounding perceived and collective social norms found among male soldiers that have been connected to sexual aggression. These discussions are used to promote bystander intervention among participants and help identify the prosocial attitudes that may be more common than previously perceived.

SUMMARY:
The proposed project will provide data concerning dating and sexual interactions that occur on Fort Bragg, North Carolina, in addition to piloting a sexual assault prevention program through the use of social norms and bystander intervention concepts. The investigators will be able to use data and feedback gained from this research to help reduce rates of sexual assault in the military by providing a sexual assault prevention program tailored to at risk male Soldiers that can be disseminated across military posts.

DETAILED DESCRIPTION:
Research has shown that one beneficial preliminary step to sexual assault prevention is the examination of a population's social norms pertaining to sex, dating, and alcohol- use. Studies show that the social norms surrounding these behaviors can be risk factors that increase the likelihood that certain high-risk men will perpetrate sexual assault.

Among college-age men, research on social norms has been used to inform the development of a sexual assault prevention program that positively impacts high-risk men. A hallmark of this approach is its exploration of the climate of a given population with regard to sex, dating and alcohol-use, and its use of data gathered to inform the development of a sexual assault program. Researchers have yet to study the effectiveness of this approach in the U.S. Army.

It has been well documented that sexual assault in the Army carries a significant threat to the readiness of the force. As such, the Army continues to make strong and laudable efforts to reduce sexual assault. However, there remains a need to better understand how young at-risk men behave in the social situations where sexual assault can occur and what they subjectively believe about these behaviors in order to effectively reduce perpetration.

In order to fill this gap, the investigators propose to implement a sexual assault prevention program by using social norms and bystander approach concepts via surveys, interviews and group workshops. The data and feedback from this research have the potential to produce insight that could help leaders and the investigators more effectively promote health in male Soldiers' dating and sexual relationships.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Active-duty Soldier (Active-duty Army, Activated Reservist or National Guardsmen) at Fort Bragg, NC
* Between the ages of 18 and 26; usage of "18-26" means at least 18 years of age but less than 27 years of age
* Reported having engaged in oral, vaginal, or anal sex within previous 4 months
* Able to speak and comprehend English sufficiently to complete the study procedures
* Indicate at risk-drinking via an AUDIT-C score >4

Exclusion Criteria:

* Screen positive for alcohol withdrawal on the ASWC (score of > 23)
* Report or indicate suicidal or homicidal ideation

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male, Active duty Soldier (Active-duty Army, Activated Reservist and National Guardsmen) at Fort Bragg, NC
Enrollment: 82 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility and impact of a sexual assault prevention program on active duty male Army Service members, Activated Reservists, and Activated National Guardsmen as assessed by surveys. | 12 months
  The purpose of the surveys is to collect quantitative data to determine the relative impact of the intervention program on participants' sexual behaviors and alcohol use.
The feasibility and impact of a sexual assault prevention program on active duty male Army Service members, Activated Reservists, and Activated National Guardsmen as assessed by individual Motivation Interviews. | 12 months
  These Motivational Interviews aim to promote change through open-ended questions, affirmations, and reflections.
The feasibility and impact of a sexual assault prevention program on active duty male Army Service members, Activated Reservists, and Activated National Guardsmen as assessed by group workshops. | 12 months
  The purpose of the group workshops is to create discussions surrounding perceived and collective social norms found among male soldiers that have been connected to sexual aggression. These discussions are used to promote bystander intervention among participants and help identify the attitudes that may be more common than previously perceived.

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Berry-Caban, PhD, Principal Investigator — Womack Army Medical Center
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be housed on a secure server in the Department of Clinical Investigation at Womack Army Medical Center. All information will be treated as confidential material and access will be restricted to research staff.